Consent Version: 03/10/2020 IRB Number: 8251

#### **Consent Form**

### **University of Oklahoma Health Sciences Center (OUHSC)**

Neuromodulation of Inflammation to Treat Heart Failure with Preserved Ejection Fraction (TIN HF)

Sponsor: National Institutes of Health

Stavros Stavrakis, MD, PhD

This is a clinical trial (a type of research study). Clinical trials include only patients who choose to take part in them. Please take your time to make your decision. Discuss this with your family and friends.

## Why Have I Been Asked To Participate In This Study?

You are being asked to take part in this study because you have been diagnosed as having heart failure with a preserved ejection fraction (meaning, your heart muscle contracts normally but the ventricles do not relax as they should).

## Why Is This Study Being Done?

The purpose of this study is to find out whether electrical stimulation of the vagus nerve using a transcutaneous electrical nerve stimulation (TENS) device can improve heart dysfunction and associated inflammation.

The TENS device is a small, portable, battery-powered device. It sends low-level, electrical pulses to the nerves under the skin of your ear through an ear clip attached to the ear.

### What is the Status of the Device Involved in this Study?

The TENS device is not approved for this use by the US Food and Drug Administration, and is being used in this study as an investigational device. This device has been studied in another heart condition called atrial fibrillation and was found to be safe and well tolerated at the pulse levels used in this study.

#### **How Many People Will Take Part In The Study?**

About 72 people will take part in this at this location.

## What Is Involved In The Study?

You will have 3 study visits: baseline, 1 month, and 3 months. Each visit will last for approximately 1 hour. At the baseline visit you will be randomized to inactive or active TENS stimulation. Randomization means that you are put in a group by chance, like the





Consent Version: 02/26/2020 IRB Number: 8251

flip of a coin. A computer program at the study site will make this random assignment. Neither you nor your physician will choose or know which group you will be assigned to.

Heart dysfunction will be assessed by using an echocardiogram (ultrasound of the heart) and an electrocardiogram (EKG), as well as a 6-minute walk test. Inflammation will be assessed in a blood sample.

During your first (baseline) visit, you will be instructed on how to use the TENS device and then you will be asked to use the device by yourself at home for 1 hour daily for 3 months. You will be asked to keep a daily diary with the time and duration of the TENS application, amplitude settings and any comments related to each daily session. The diary will take approximately less than 5 minutes to complete.

During the baseline and 3 month visits you will have the following at each visit: a medical history taken and physical examination, any cardiovascular events will be recorded, asked to complete a questionnaire, an echocardiogram, about 10cc (2) teaspoons) of blood drawn, a 6- minute walk test and a 5 minute and 10 second EKG.

During the 1 month visit you will be interviewed by the research coordinator to address any issues with the use of the TENS device at home, and to make sure that you are using it correctly.

At the end of the study, you will be asked to return the TENS device back to the study doctor.

## **How Long Will I Be In The Study?**

You will be in the study for 3 months of follow up. You can stop participating in this study at any time. However, if you decide to stop participating in the study, we encourage you to talk to the researcher first.

There may be anticipated circumstances under which your participation may be terminated by the investigator without regard to your consent.

- He/She feels that it is in your medical best interest.
- You fail to follow study requirements.

#### What Are The Risks of The Study?

Use of the TENS device for electrical ear stimulation therapy may involve risks that are currently unforeseeable.

The TENS device has been found to be very safe and well tolerated when used correctly. You could experience some minor side effects: some numbness, tingling sensation, or mild skin irritation at the site of application on your ear, skin redness and pressure marks at the site of stimulation, painful stimulation, dysesthesia (abnormal skin sensation), dizziness, mild shortness of breath and headaches. More significant side effects like heart arrhythmias are extremely rare.



Consent Version: 02/26/2020 IRB Number: 8251

The risks of a blood draw include fainting, mild pain, local irritation or bruising, swelling or bleeding. In rare cases the area where the needle is inserted can also become infected or nerves may be damaged, inducing long-lasting abnormal sensations (paresthesia), impaired sensation of touch, and persistent pain.

#### **Are There Benefits to Taking Part in The Study?**

If you agree to take part in this study, there may or may not be direct medical benefit to you. We hope that the information learned from this study will benefit other patients with this disease in the future.

### What Other Options Are There?

You may choose not to participate in the study. Please talk to your regular doctor about these and other options

## What about Confidentiality?

Efforts will be made to keep your personal information confidential. You will not be identifiable by name or description in any reports or publications about this study. We cannot guarantee absolute confidentiality. Your personal information may be disclosed if required by law. You will be asked to sign a separate authorization form for use or sharing of your protected health information.

There are organizations outside the OUHSC that may inspect and/or copy your research records for quality assurance and data analysis. These organizations include the US Food & Drug Administration and other regulatory agencies. The OUHSC Human Research Participant Program office, the OUHSC Institutional Review Board, and the OUHSC Office of Compliance may also inspect and/or copy your research records for these purposes.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. However, this website will not include information that can identify you. At most, the website will include a summary of the study and results. You can search this website at any time.

#### **Certificate of Confidentiality:**

To help protect your privacy, this research is covered by a Certificate of Confidentiality from the National Institutes of Health. This Certificate means that the researchers cannot be forced (for example by court subpoena) to share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate cannot be used to resist a demand for information from personnel of the U.S. government that is used for checking or evaluating federally-funded projects or for information that must be disclosed in order to meet the requirements of the US Food and Drug Administration.





Consent Version: 02/26/2020 IRB Number: 8251

The protection offered by the Certificate of Confidentiality does not prevent us from being required by applicable state law to report information about suspected or known sexual, physical, or other abuse of a child or older person, or a subject's threats of violence to self or others. If any member of the research team is given such information, he or she will be required to make a report to the appropriate authorities.

The Certificate, however, does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information. This means that you and your family should actively protect your own privacy.

#### What Are the Costs?

There is no cost to you if you participate in this study. The use of the TENS device, study visits, lab work, EKGs, 6-minute walk test, and echocardiogram will be provided at no charge to you or your insurance company.

### Will I Be Paid For Participating in This Study?

You will receive a \$40 gift card for each study visit.

# What if I am Injured or Become III While Participating in this Study?

In the case of injury or illness resulting from this study, emergency medical treatment is available. However, you and/or your insurance company will be responsible for the cost of the treatment. No funds have been set aside by The University of Oklahoma Health Sciences Center, the National Institutes of Health or the study doctor to compensate you in the event of injury.

#### What Are My Rights As a Participant?

Taking part in this study is voluntary. You may choose not to participate. Refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled. If you agree to participate and then decide against it, you can withdraw for any reason and leave the study at any time. Please be sure to discuss leaving the study with the principal investigator or your regular doctor. You may discontinue your participation at any time without penalty or loss of benefits to which you are otherwise entitled.

We will provide you with any significant new findings developed during the course of the research that may affect your health, welfare, or willingness to continue your participation in this study.

You have the right to access the medical information that has been collected about you as a part of this research study. However, you may not have access to this medical information until the entire research study has completely finished. You consent to this temporary restriction.



Consent Version: 02/26/2020 IRB Number: 8251

### Whom Do I Call If I have Questions or Problems?

If you have questions, concerns, or complaints about the study or have a research-related injury, Dr. Stavros Stavrakis can be reached 24 hours a day, seven days a week at the following number: 405-271-9696.

If you cannot reach the Investigator or wish to speak to someone other than the investigator, contact the OUHSC Director, Office of Human Research Participant Protection, at 405-271-2045.

For questions about your rights as a research participant, contact the OUHSC Director, Office of Human Research Participant Protection at 405-271-2045.

#### **Signature:**

By signing this form, you are agreeing to participate in this research study under the conditions described. You have not given up any of your legal rights or released any individual or entity from liability for negligence. You have been given an opportunity to ask questions. You will be given a copy of this consent document.

| I agree to participate in this study: | | |
|------------------------------------------|--------------|------|
| PARTICIPANT SIGNATURE (age ≥18) | Printed Name | Date |
| SIGNATURE OF PERSON<br>OBTAINING CONSENT | Printed Name | Date |

IRB Office Version Date: 09/21/2016

